CLINICAL TRIAL: NCT02956785
Title: What After the First Propess. A Randomised Comparative Prospective Study
Brief Title: What After the First Propess
Acronym: PRODUCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit more women because of the COVID-19 and staffing/resources issues
Sponsor: South Warwickshire NHS Foundation Trust (Other)
Collaborators: Medicem International (Unknown); Walsall Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, Amr Farag, Consultant Obstetrician and Gynaecologist, Walsall Healthcare NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202984
Record Dates: First submitted 2016-10-29; First posted 2016-11-07 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Induction of Labor
Keywords: Propess
MeSH Terms: interventions — Dinoprostone; KLK15 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Extension of propess+/-second propess (Active Comparator): Women will have the initial slow-release Dinoprostone pessary left in place for six more hours (total of 30 hours in place) then removed followed by vaginal assessment 48 hours after the start of labour induction and insertion of a second slow-release pessary if required
  Interventions: Drug: 10 mg Dinoprostone; CTS, UK
- Prostin (Active Comparator): Women will have the initial slow-release Dinoprostone pessary removed followed by insertion of quick-release Dinoprostone tablet (Prostin® 3 mg Dinoprostone vaginal tablet; Pfizer, UK) high in the posterior vaginal fornix immediately after removal of the slow-release pessary. The tablet will be left for 6 hours followed by vaginal reassessment and insertion of a second tablet if ARM is still not achievable.
  Interventions: Drug: 3 mg Dinoprostone vaginal tablet; Pfizer, UK
- Dilapan-S (Active Comparator): Women will have the initial slow-release Dinoprostone pessary removed followed by insertion of 1-5 Osmotic cervical rods (Dilapan-S® Aquacryl hydrogel rod; HPSRx Enterprises, USA) by a senior obstetrician or a midwife into the cervical canal, immediately after removal of the slow-release pessary using a vaginal speculum and a holder. The rods will be left for 12-24 hours.
  Interventions: Drug: Aquacryl hydrogel rod; HPSRx Enterprises, USA

INTERVENTIONS:
Drug: 10 mg Dinoprostone; CTS, UK
  Other Names: Propess
  Arms: Extension of propess+/-second propess
Drug: 3 mg Dinoprostone vaginal tablet; Pfizer, UK
  Other Names: Prostin
  Arms: Prostin
Drug: Aquacryl hydrogel rod; HPSRx Enterprises, USA
  Other Names: Dilapan-S
  Arms: Dilapan-S

SUMMARY:
The aim of this study is to compare three different regimens for continuation of induction of labor after no spontaneous or artificial rupture of membranes could be achieved after first 24 hours post-insertion of Dinoprostone

DETAILED DESCRIPTION:
This randomized study will be carried out at delivery suite in Warwick Hospital after eligible women have been informed of the study when booked for induction of labor and provided with the study information leaflet

When attending for induction of labor on delivery suite, an informed consent will be obtained then all women will have a cardiotocogram (CTG) performed initially and will be assessed by vaginal examination and Bishop score recorded at insertion of first slow-release pessary (Propess®10 mg Dinoprostone; CTS, UK), which will be inserted high into the posterior vaginal fornix. Assessment and insertion of pessary will be done by an experienced obstetrician or a senior midwife

All women will be given the required care and support as per the local protocols and guidelines

Women will be excluded from the study within the first 24 hours of induction of labor in the following conditions:

* Women with abnormal or non-reassuring CTG needing intervention.
* Women needing tocolytic use.
* Women needing removal of the Dinoprostone pessary.
* Women needing emergency Caesarean section.
* If spontaneous rupture of membranes occurs.
* If artificial rupture of membranes is achievable after the first 24 hours of induction of labor (Bishop score 5 or more)
* If woman withdraws her consent to continue as a part of the study.

After 24 hours from insertion of the first Dinoprostone pessary, women will be reassessed and a total of 330 women with Bishop score less than 7, will be randomly assigned to one of three intervention groups by a pre-formed computer-generated random list and randomization put in sealed opaque envelopes kept in a locked secure area on delivery suite.

Intervention groups will be as follows:

Group 1 (110 women):

Women will have the initial slow-release Dinoprostone pessary left in place for six more hours (total of 30 hours in place) then removed followed by vaginal assessment 48 hours after the start of labour induction and insertion of a second slow-release pessary if required (Currently Propess® is not licensed to be repeated as a second dose. However, there is a consensus that, the dose may be repeated after a consultant review and an informed verbal consent as per SWH 00190 Induction and Augmentation of the First and Second Stage of Labour Management Guideline, 2012).

Group 2 (110 women):

Women will have the initial slow-release Dinoprostone pessary removed followed by insertion of quick-release Dinoprostone tablet (Prostin® 3 mg Dinoprostone vaginal tablet; Pfizer, UK) high in the posterior vaginal fornix immediately after removal of the slow-release pessary. The tablet will be left for 6 hours followed by vaginal reassessment and insertion of a second tablet if ARM is still not achievable.

Group 3 (110 women):

Women will have the initial slow-release Dinoprostone pessary removed followed by insertion of 1-5 Osmotic cervical rods (Dilapan-S® Aquacryl hydrogel rod; HPSRx Enterprises, USA) by a senior obstetrician or a midwife into the cervical canal, immediately after removal of the slow-release pessary using a vaginal speculum and a holder. The rods will be left for 12-24 hours.

For all participants, after achieving spontaneous or artificial rupture of membranes, the local protocol for intrapartum care will be followed and after delivery, the women will be asked to fill in a patient's satisfaction questionnaire about the process of induction, care given and being a part of the study

ELIGIBILITY:
Inclusion Criteria:

* Women booked for induction of labor at 37 to 42 weeks gestation
* Viable singleton pregnancy.
* Cephalic presentation.
* Intact membranes.
* No previous Caesarean section.
* No antenatal fetal concerns (Fetal growth restriction (FGR), small for gestational age (SGA), impaired Doppler, oligohydramnios, non-reassuring/abnormal CTG).

Exclusion Criteria:

* Pregnancy less than completed 37 weeks or more than 42 weeks.
* Multiple pregnancy.
* Intrauterine fetal death.
* Non-cephalic presentation.
* Pre-labor rupture of membranes
* Previous one or more Caesarean sections.
* Antenatal concerns regarding fetal well-being (FGR, SGA, impaired Doppler, oligohydramnios, non-reassuring/abnormal CTG).
* Non-reassuring or abnormal CTG on admission to labor ward

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Rate of achieving spontaneous or artificial rupture of membranes | 12 months
  percentage of women who will have spontaneous or artificial rupture of membranes

SECONDARY OUTCOMES:
Time interval needed from start of induction of labor to achieve spontaneous or artificial rupture of membranes | 12 months
  The time frame is 6 months from the onset of the study till assessing the results, doing the analysis and presenting.
  But, the time interval stated as an outcome here is the period of time elapsing from starting induction of labour and rupturing the membranes whether spontaneous or artificial
Rate of hyperstimulation (contractions more than 5 in 10 minutes or each contraction lasting more than 90 seconds) | 12 months
  percentage of women who will develop uterine hyperstimulation
Rate of abnormal CTG changes needing intervention | 12 months
  percentage of women with non-reassuring or abnormal CTG that need intervention
Rate of need for tocolysis | 12 months
  percentage of women who need tocolysis to treat hyperstimulation
Rate of emergency Caesarean section | 12 months
  percentage of women who need Caesarean section for fetal distress or failed induction/progress of labour
Grades of Caesarean sections | 12 months
  percentage of each of grade 1,2 and 3 Caesarean sections among each group
Women's satisfaction with the method of induction used | 12 months
  scoring system based on women's questionnaire formed of 3 questions with a score of 3 to 15. In addition, evaluation of pain score out of 10

CONTACTS AND LOCATIONS:
Overall Officials: Amr H Farag, Consultant, Principal Investigator — Walsall Healthcare NHS Trust
Locations (1):
- Walsall Healthcare NHS Trust, Walsall, United Kingdom